CLINICAL TRIAL: NCT02147483
Title: Mindfulness-Based Relapse Prevention and Stress Reactivity in Alcohol Dependent Individuals: A Pilot Study
Brief Title: Mindfulness-Based Relapse Prevention for Alcohol Use Disorders in Remission
Acronym: MBRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jennifer Kim Penberthy, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16363
Record Dates: First submitted 2013-11-14; First posted 2014-05-26 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Alcohol Use Disorders
Keywords: Mindfulness; Alcohol use disorders
MeSH Terms: conditions — Alcoholism | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as usual (Active Comparator): Treatment as usual as prescribed by clinician.
  Interventions: Behavioral: Treatment as usual
- Mindfulness Based Relapse Prevention (Experimental): Mindfulness based relapse prevention will be provided in eight in person sessions to prevent alcohol use.
  Interventions: Behavioral: Mindfulness Based Relapse Prevention

INTERVENTIONS:
Behavioral: Mindfulness Based Relapse Prevention — Mindfulness based relapse prevention therapy provided over eight sessions in person to prevent alcohol relapse.
  Arms: Mindfulness Based Relapse Prevention
Behavioral: Treatment as usual — Treatment usually provided by clinician
  Arms: Treatment as usual

SUMMARY:
We propose to conduct a pilot study that will examine the utility and mechanisms of Mindfulness-Based Relapse Prevention in reducing alcohol consumption, relapse rates, and physiological arousal to stress in adults 21 years of age and older who have met DSM-IV-TR diagnostic criteria for alcohol dependence within the past year but have abstained from drinking for the last thirty days. MBRP is designed to improve one's ability to self-regulate emotions, thoughts and physical states, thus reducing the need to alleviate associated discomfort through substance use. Participants assigned to the intervention group will receive an 8-week training course of MBRP over a period of nine weeks; participants assigned to the Treatment As Usual (TAU) group will continue treatment as usual, which includes utilizing their own effective strategies to refrain from alcohol use. All participants will be assessed for pretreatment severity of psychological abuse/trauma as well as pre and posttreatment psychosocial functioning (e.g., alcohol consumption, symptoms of depression and anxiety, emotion regulation/coping). The outcome of treatment will be evaluated using a) Timeline Followback drinking data and b) self-report ratings of acquisition of MBRP skills (e.g., state/trait mindfulness, acceptance and awareness, and perceived stress) and depressive and anxiety symptom severity. We hypothesize that participants who receive MBRP training will demonstrate greater acceptance and awareness, reduced cravings, and have a lower likelihood of relapse than participants in the TAU group. It is also expected that MBRP participants will demonstrate greater improvements on psychological measures of depression, anxiety, emotion regulation and coping, and show less perceived stress and physiological arousal to stress compared to TAU participants. Finally, little is known about which types of individuals are most likely to benefit from MBRP. Thus, secondary analyses will help to clarify for whom MBRP may be most effective.

DETAILED DESCRIPTION:
Stress exposure increases psychological and physiological arousal and can lead to negative health outcomes. An impaired ability to self-regulate in response to stress contributes to the development of alcohol use disorders and relapse. Mindfulness, a state of present-focused attention and awareness, can be systematically learned through meditative practice to improve self-regulation of emotional, physiological and behavioral responses to stress. Mindfulness meditation further facilitates a balance of mind and body thereby increasing one's ability to respond proactively and effectively to daily events. Research evidence suggests a strong association between mindfulness and positive indicators of well-being which include reductions in fear, anxiety, anger, and better physiological recovery from stress.

Given the importance of self-regulation in the development and progression of alcohol use disorders and relapse, a new approach to substance use treatment, Mindfulness-Based Relapse Prevention (MBRP), was developed. Traditionally, MBRP is an eight-week outpatient treatment program, which integrates core aspects of Relapse Prevention (RP) practices with practices adapted from Mindfulness-Based Stress Reduction (MBSR) and Mindfulness-Based Cognitive Therapy. The mindfulness practices in MBRP are designed to increase acceptance and tolerance of negative emotions, thoughts and physical states thus reducing the need to alleviate associated discomfort through substance use. MBRP also focuses on increasing awareness of triggers and developing more effective coping behaviors in high-risk situations. Among adults with substance use disorders, MBRP has been found to lead to significantly lower rates of substance use, greater decreases in cravings and greater increases in acceptance and acting with awareness than treatment as usual. MBRP has also been found to facilitate more effective coping and self-regulation of negative emotions during early abstinence.

While research indicates that MBRP is effective in reducing substance use relapse, only preliminary research has examined the influence of MBRP on the physiological mechanisms involved in emotion regulation after exposure to stress. Examining these physiological mechanisms is essential because the central and autonomic nervous systems work together to coordinate the self-regulation of attention, cognition and emotion when stressful cues are encountered, such as when a substance dependent individual is exposed to stressful and/or substance related stimuli. Heart rate variability (HRV) is generally seen as an index of emotion regulation. High frequency HRV reflects parasympathetic activation of the autonomic nervous system and the body's ability to exert cognitive control over attention and emotional responding. Higher levels of HRV are associated with greater emotional and behavioral flexibility, and tend to be associated with better mental and physical health outcomes. In contrast, lower levels of HRV are associated with a wide range of medical and psychiatric disorders, including acute and chronic alcohol ingestion, anxiety and depression. Among alcohol dependent individuals, mindfulness training has been found to increase HRV and lower subjective levels of psychological distress in response to stressful cues in the short-term. The proposed study will be the first to examine the long-term effects of MBRP on HRV and self-reported psychological/behavioral functioning. The results will provide a better understanding of the interplay between the psychological and physical mechanisms involved in relapse and help determine whether MBRP has lasting psychological and physiological benefits. In other words, assessing both the psychological and physiological effects of MBRP will provide a more accurate and comprehensive understanding of how mindfulness aids in promoting self-regulation and relapse prevention. Finally, little is known about which types of individuals are most likely to benefit from MBRP. It is necessary to examine individual characteristics (i.e., baseline levels of HRV, trait mindfulness, substance use, anxiety, depression) to determine which characteristics are associated with positive treatment outcomes in both the short and long-term. This knowledge will enable more efficient and effective delivery of the MBRP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who have given written informed consent
* 21 years of age or older
* DSM-IV-TR diagnosis of alcohol dependence within the last year, but have abstained from drinking for the last thirty days
* Literate in English and able to read, understand, and complete the rating scales and questionnaires accurately, follow instructions, and make use of mindfulness techniques
* Express a wish to remain abstinent from drinking
* Willingness to participate in mindfulness techniques
* Able to attend all clinic visits without interruption

Exclusion Criteria:

* Any current Axis I DSM-IV-TR psychiatric disorder other than alcohol or nicotine dependence that, in the clinician's opinion, warrants treatment or would preclude safe participation in the protocol, including, but not limited to: psychosis, schizophrenia, dementia, schizotypal personality disorder, borderline personality disorder, bipolar disorder, primary diagnosis of eating disorder, or chronic suicidality or homicidality
* Current use of Antabuse (Disulfiram) to pharmacologically treat alcohol dependence
* Serious medical comorbidity requiring medical intervention or close supervision, including a history of dangerous symptoms of withdrawal from alcohol (e.g., seizures), pacemakers, heart transplant, severe arrhythmias, or active atrial fibrillation
* Suicide attempt in the last thirty days
* Gross neurological disease
* Mental retardation, which will be assessed by the PI, postdoctoral fellows, and doctoral students in clinical psychology)
* Minors below the legal drinking age will not be included.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2016-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Mindfulness levels | up to 4 months post treatment
  Difference scores on mindfulness scales (session 04 minus baseline, session 08 minus baseline, two-month follow-up minus baseline, four-month follow-up minus baseline) will be calculated. 2 group (intervention, TAU) x 5 interval (baseline, session 04, session 08, two-months follow-up, four-months follow-up) repeated measures analyses of variance (ANOVAs) will be conducted.

SECONDARY OUTCOMES:
cravings; symptoms of depression, anxiety, and perceived stress; obsessive thoughts of alcohol/compulsive drinking | up to 4 months post treatment
  Difference scores (session 04 minus baseline, session 08 minus baseline, two-month follow-up minus baseline, four-month follow-up minus baseline) will be calculated for cravings, symptoms of depression, anxiety, perceived stress, obsessive thoughts of alcohol/compulsive drinking. To test hypotheses 1, 2, and 3, 2 group (intervention, TAU) x 5 interval (baseline, session 04, session 08, two-months follow-up, four-months follow-up) repeated measures analyses of variance (ANOVAs) will be conducted.

OTHER OUTCOMES:
drinking behavior | up to 4 months post treatment
  Difference scores (session 04 minus baseline, session 08 minus baseline, two-month follow-up minus baseline, four-month follow-up minus baseline) will be calculated for total drinks. 2 group (intervention, TAU) x 5 interval (baseline, session 04, session 08, two-months follow-up, four-months follow-up) repeated measures analyses of variance (ANOVAs) will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Penberthy, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia School of Medicine, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No